CLINICAL TRIAL: NCT03778593
Title: Phase II Trial of Modified FOLFIRINOX in Patients With Metastatic Biliary Tract Cancer After Failure of Gemcitabine/Cisplatin Chemotherapy
Brief Title: FOLFIRINOX for 2nd-line Treatment of BTC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A University Hospital (Other)
Responsible Party: Principal Investigator, Sung Yong Oh, Associate Professor, Dong-A University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GF BTC-2018
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Biliary Tract Cancer
Keywords: biliary tract carcinoma; 5-FU; Irinotecan; oxaliplatin
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Fluorouracil; Leucovorin; Irinotecan; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: mFOLFIRINOX (5-FU, Irinotecan, oxaliplatin, Leucovorin)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mFOLFIRINOX (Experimental): D1 Oxaliplatin 65 mg/m2 + 5% dextrose water (5DW) 200 mL mix IV over 2 hours followed by, D1 Leucovorin 400 mg/m2 + 5DW 200 ml mix IV over 2 hours D1 Irinotecan 135 mg/m2 + 5DW 500 mL mix IV over 2 hours (concurrent with the leucovorin infusion) D1-2 5-Fluorouracil 1000 mg/m2 + 5DW 1 liter (1L) continuous IV over 23 hours repeat every 2 weeks
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Irinotecan; Drug: Oxaliplatin; Drug: 5% dextrose water

INTERVENTIONS:
Drug: 5-Fluorouracil — D1-2 5-Fluorouracil 1000 mg/m2 + 5DW 1L continuous IV over 23 hours q 2 weeks
Drug: Leucovorin — D1 Leucovorin 400 mg/m2 + 5DW 200 ml mix IV over 2 hours q 2 weeks
Drug: Irinotecan — D1 Irinotecan 135 mg/m2 + 5DW 500 mL mix IV over 2 hours (concurrent with the leucovorin infusion) q 2weeks
Drug: Oxaliplatin — D1 Oxaliplatin 65 mg/m2 + 5DW 200 mL mix IV over 2 hours q 2 weeks
Drug: 5% dextrose water — mix fluid with 5-FU, leucovorin, irinotecan, and oxaliplatin
  Other Names: 5DW

SUMMARY:
Biliary tract cancer (BTC) is rare in the West, but it is relatively high in Asia, including Korea. Currently used as the standard primary treatment in metastatic or locally advanced BTC is gemcitabine/platinum combination chemotherapy.There is no standard secondary chemotherapy recognized after the failure of the gemcitabine/platinum first line treatment. The investigators try to evaluate role of 5-FU, leucovorin, irinotecan, and oxaliplatin combination chemotherapy (FOLFIRINOX) for the patients who progressed after gemcitabine/cisplatin first line chemotherapy.

DETAILED DESCRIPTION:
<Biliary tract cancer> Biliary tract cancer (BTC) is a common term for malignant tumors that occur in gallbladder and bile duct, the path in which bile is released. According to the anatomical location, biliary tract cancer is divided into intrahepatic cholangiocarcinoma and extrahepatic cholangiocarcinoma, and extrahepatic cholangiocarcinoma is classified as perihilar cholangiocarcinoma and distal cholangiocarcinoma. Biliary tract cancer is rare in the West, but it is relatively high in Asia, including Korea. Biliary tract cancer occurs annually in Korea, accounting for about 5,600 cases, 2.4 percent of the total cancer, and ranks sixth in deaths from cancer. Biliary tract cancer is a type of cancer that is difficult to treat because most patients are diagnosed with progressive diseases that cannot be operated. Only about a quarter of patients are diagnosed with surgical-ready conditions as a treatment where full surgical operation can be expected to complete, but the five-year survival rate for operation is poor at 8-44% due to a high recurrence after surgery.

<Metastatic or relapsed biliary tract cancer treatment> Chemotherapy is the main treatment in BTC, which is relapsed or metastatic status. 5- Fluorouracil (5-FU)-based treatment has been shown to improve the survival period for pancreatic and bile cancer patients compared to the optimal supportive care (5-FU/leucovorin ± etoposide 6.0 vs. 2.5 months, p <0.01). Also, chemotherapy helped maintain the quality of life. The improvement in quality of life over a period of at least four months showed a significant difference compared to 10% in the group that received only optimal supportive care for 36% of the chemotherapy group. (p < 0.01). Currently used as the standard primary treatment in metastatic or locally advanced BTC is gemcitabine/platinum combination chemotherapy. In a large phase III study, Gemcitabine/cisplatin significantly improved the median value of the progressive free survival (PFS) period from 5.0 months to 8.0 months, and the overall survival (OS) period from 8.1 months to 11.7 months, compared to the gemcitabine alone. If Cisplatin is not available, oxaliplatin can be considered as a merger with gemcitabine. The Gemcitabine/oxaliplatin regimen reported in the phase II and phase III studies PFS was 4.2-5.5 months, median for the OS period was 9.5-12.4 months.

<Salvage treatment of biliary tract cancer> To date, there is no standard secondary chemotherapy recognized after the failure of the gemcitabine/platinum primary treatment. Since BTC usually occurs at an advanced age and shows a low frequency of occurrence in the West, there are practical limitations to conducting large-scale clinical research. So far, there is no large three-phase study proving the benefits of secondary chemotherapy after the failure of gemcitabine/platinum chemotherapy. Implementation of secondary chemotherapy in actual clinicians is known to vary from country to country, depending on the medical judgment of the responsible clinician. In a large-scale retrospective study by the Association des Gastro-Enterologies Oncology (AGEO) group in France, 32.5% of the patients were treated with second line therapy, and 75% of the patients were reported in Japan. A retrospective study and a two-phase study and systematic literature review suggest that there will be a benefit from the treatment if second line treatment is selected for patients whose general health is relatively well maintained. Results of single or combination therapy using drugs such as Irinotecan, oxaliplatin, 5-FU, S-1, and capecitabine were reported in phase II and retrospective studies, yielding an average of 3.2 months of PFS, 7.7% of mean response rate, and 7.2 months of OS.

The 5-FU/leucovorin/irinotecan (FOLFIRI) therapy, along with the capecitabine/irinotecan therapy, is reported as the most commonly used secondary chemotherapy in the AGEO group in France. A treatment strategy for continuous use of FOLFIRI as a secondary treatment after the failure of Gemcitabine/oxaliplatin showed the median value for OS period of 21.9 months, and the median value for the PFS period. The PFS and OS due to the FOLFIRI was found to be 3.2 months and 8.4 months, respectively. On the other hand, the FOLFOX therapy, which combines oxaliplatin with 5-FU, showed a response rate of 21.6 % when administered as a secondary treatment after the failure of gemcitabine/cisplatin, and a median PFS of 3.1 months. A phase III study is currently underway that compares the administration of FOLFOX as a secondary treatment with the optimum support. In Korea, there is a problem with the standard reimbursement for applying to drugs prescribed to cancer patients, and in particular, cancer drugs that can be used as secondary therapy in metastatic BTC patients are limited. There is a need to improve the prognosis of BTC patients by expanding the use of various drugs that have been proven through external clinical research.

<5-FU, leucovorin, irinotecan, and oxaliplatin combination chemotherapy (FOLFIRINOX) regimen for other cancer of BTC> In a pre-clinical experiment, oxaliplatin and irinotecan have synergistic effects and are known to have relatively no overlap of toxic effects among, 5-FU, leucovorin, irinotecan, and oxaliplatin. The combination treatment of 5-FU/leukovorin/irinotecan/oxaliplatin (FOLFIRINOX) had a high therapeutic effect on progressive pancreatic cancer and colon cancer. In a phase III study comparing FOLFIRINOX and gemcitabine as a first line treatment in metastatic pancreatic cancer, the objective response rate (32 vs. 9%), PFS (6.4 vs. 3.3 months) and OS (11.1 vs. 6.8 months) were significantly higher in FOLFIRINOX. On the other hand, treatment-related toxicities, with a grade 3/4 of neutropenia (46 vs. 21%), febrile neutropenia (5.4 vs. 1.2%), thrombocytopenia (9.1 vs. 3.6%), sensory neuropathy (9 vs. 0%), vomiting (23 vs. 18%), and diarrhea (113 vs. 2%) were more common in FOLFIRINOX. In a phase III study comparing the 5-FU/leukovorin/irinotecan/oxaliplatin(FORFOXRI) and the 5-FU/leukovorin/irinotecan(FORFIRI) as a first line treatment in metastatic colorectal cancer, the FORFOXRI group was objective response (66 vs. 41 %), the PFS (9.8 vs. 6.9 months) and the OS (2.6 vs. 16.7 months) showed significant improvements. In pancreatic cancer, FOLFIRINOX was a treatment that was limited in patients with good general condition due to its high level of toxicity, including neutropenia, but the dose-reduction proved to be applied not only as a primary treatment but also as a secondary treatment. In a phase II study of pancreatic cancer patients in China, there was a 29% of grade 3/4 neutropenia were reported due to the treatment of modified FOLFIRINOX using oxaliplatin 68 mg/m2, irinotecan 135 mg/m2, and 5-FU injection of 2,400 mg/m2 for 46 hours, and there was no increase in mortality and febrile neutropenia. Other major grade 3 or higher toxicity levels showed improved safety profiles with thrombocytopenia (4.8%), anemia (8.1%), infection (4.8%), and elevated liver enzyme (14.5%).

<Rationale of this trial>

As a 2nd line treatment for metastatic BTC the assessment of modified FOLFIRINOX is supported by:

* The prognosis for metastatic BTC, which fails first line therapy, is poor and has no standardized treatment. Therefore, better treatment modalities are required to improve the survival of patients who no longer respond to first line treatment and to maintain the quality of life.
* Treatments that use irinotecan or oxaliplatin as secondary therapy for metastatic BTC have been shown in retrospective and phase II studies and are actually used in clinical practice of other countries.
* Oxaliplatin and irinotecan have synergistic effects and the FOLFIRINOX therapy, which uses both drugs together in 5-FU/leucovorin, has been shown to increase efficacy in pancreatic and colon cancer.
* The modified FOLFIRINOX, which was used with reduced dosage, indicates an acceptable toxic profile while maintaining its efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed BTC (cholangiocarcinoma or gall bladder (GB) cancer) , except ampulla of Vater cancer
2. In the event that the progression of the gemcitabine/cisplatin is experienced during or after discontinuation of the first line treatment for metastatic, locally advanced or relapsed (it may be considered as a first line treatment that recurrence within six months of completion of the adjuvant or neo-adjuvant chemotherapy using gemcitabine/cisplatin)
3. Patient (or legal representative) has completed an approved consent documents that he or she will participate in the test after receiving sufficient information about the clinical trial
4. East clinical oncology group (ECOG) performance status 0-1
5. One or more measurable lesions by RECIST v1.1.
6. Appropriate organ functions; A. Liver: bilirubin ≤ 3 mg/dL, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 x ULN (in cases of liver metastasis, AST or ALT ≤ 5 x ULN) B. Kidney: An estimate of creatine clearance rate according to the Cockcroft-Gault formula (or local institution's standard method) > 30 mili-liter (mL)/min C. Hemoglobin ≥ 9 g/dL (transfusion allowed), absolute neutrophil count (ANC) ≥ 1500/μL, platelet count ≥ 75,000/μL.
7. Expected life time over 3 months.
8. Over 19 years old.
9. In case of proper bile excretion function
10. Have the will and ability to comply with the clinical trial plan during the study period, including treatment and scheduled visits and examination.
11. For pre-menopausal women and for women less than one year after the onset of menopause, serum or urine pregnancy tests shall be confirmed negative during screening.
12. For men and fertile women, the use of effective contraceptive methods should be agreed (effective contraception should be used for at least 30 days prior to the initial administration of a investigational drug, the trial period, and at least 90 days after the discontinuation of the test participation).

Exclusion Criteria:

1. ≥ 2 of prior chemotherapy for progressive BTC (except for adjuvant/neo-adjuvant chemotherapy with resting of more than six months)
2. Symptomatic or untreated brain metastasis or spinal cord compression metastasis.
3. Previous treatment using Irinotecan or oxaliplatin
4. In case of major surgery within four weeks just before registration, excluding biopsy for diagnosis
5. In case of chemotherapy or radiation therapy was received within three weeks prior to the administration of a test medication
6. Grade 2 or higher peripheral neuropathy
7. Grade 2 or higher toxicities caused by a previous cancer treatment based on NCI-CTCAE v 4.03 other than hair loss
8. A person diagnosed with another malignant tumor within the last five years. Exceptions include basal or squamous cell carcinoma of the skin or intraepithelial neoplasia (bladder, uterine cervical, colorectal, breast)
9. Pregnant or nursing woman
10. If there is a severe or uncontrolled systemic disease, active infection, active bleeding tendency or organ transplantation history (including allo-hematopoietic stem cell transplantation)
11. The following virus infection A. Known positive history for human immunodeficiency virus (Human Immunodeficiency virus, HIV) test or known acquired immunodeficiency syndrome (AIDS) B. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (positive Hepatitis B surface -Ag (+) or HCV RNA (+) if anti-HCV Ab screening test is positive)
12. If there is a known alcohol or drug abuse
13. In cases of clinically significant (i.e., active) cardiovascular disease: cerebral hemorrhage/brain infarction, myocardial infarction (pre-registration < 6 months), unstable angina, congestive heart failure (NYHA classification ≥2) or arrhythmia needed drug therapy.
14. In case of a mental state in which it is impossible to understand and provide the consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Response rate of treated participants | up to 6 months
  Rate of response including complete response and partial response by treatment. Response will be evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Progression free survival (PFS) duration of treated participants | up to 12 months
  duration measure from treatment day to progression + death events. Calculated by Kaplan-Meier survival analysis.
Overall survival (OS) duration of treated participants | up to 12 months
  duration measure from treatment day to death events. Calculated by Kaplan-Meier survival analysis.
Incidence of Treatment-Emergent Adverse Events of participants | up to 12 months
  all adverse events during treatment. Evaluated with National Cancer Institute(NCI)-] Common Terminology Criteria for Adverse Events (CTCAE) v4.03

OTHER OUTCOMES:
EORTC -QoL-C30 | up to 12 months
  Evaluate patients' life quality evaluation during treatment every 2 months with questionaires.
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (EORTC QOL-C30) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Oh, M.D., Principal Investigator — Dong-A University Hospital
Locations (1):
- Dong-A University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No